CLINICAL TRIAL: NCT03937830
Title: A Phase II Study of Combined Treatment of Durvalumab, Bevacizumab, Tremelimumab and Transarterial Chemoembolization (TACE) in Subjects With Hepatocellular Carcinoma (HCC) or Biliary Tract Carcinoma (BTC)
Brief Title: Combined Treatment of Durvalumab, Bevacizumab, Tremelimumab and Transarterial Chemoembolization (TACE) in Subjects With Hepatocellular Carcinoma or Biliary Tract Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190094; 19-C-0094
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-21

CONDITIONS: Hepatocellular Cancer; Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma
Keywords: Immune Checkpoint Blockade; Combined Treatment; Immunotherapy; Anti-Tumor Immunity; Inhibition of the Blood Vessels Surrounding a Tumor
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — durvalumab; Bevacizumab; tremelimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Arm 1 (Experimental): Durvalumab, bevacizumab and tremelimumab
  Interventions: Drug: durvalumab; Drug: bevacizumab; Drug: Tremelimumab
- 2/Arm 2 (Experimental): Durvalumab, bevacizumab, tremelimumab and TACE
  Interventions: Drug: durvalumab; Drug: Doxorubicin-Eluting Beads; Procedure: TACE; Drug: bevacizumab; Drug: Tremelimumab
- 3/Arm 3 (Experimental): Durvalumab, low-dose bevacizumab, and tremelimumab
  Interventions: Drug: durvalumab; Drug: bevacizumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: durvalumab — 1,150 mg flat dose every 21 days, starting on day 1 of cycle 1
Drug: Doxorubicin-Eluting Beads — used for TACE (only in patients with HCC BCLC stage B)
  Arms: 2/Arm 2
Procedure: TACE — TACE with Doxorubicin-Eluting Beads (only in patients with HCC BCLC stage B) on Cycle 2. More TACE can be done if clinically necessary.
  Arms: 2/Arm 2
Drug: bevacizumab — 7.5 mg/kg dose every 21 days, starting on day 1 of cycle 2
Drug: Tremelimumab — 300, 150 or 75 mg once on day 1 of cycle 1

SUMMARY:
Background:

Hepatocellular carcinoma (HCC) is the fifth most common cancer in the world. Most people with advanced HCC survive an average of 6 to 9 months. Researchers are evaluating a combination of treatment drugs to delay the progression of HCC; aiming to help people with HCC live longer.

Objective:

To study the 6-month progression-free survival in people with advanced HCC treated with bevacizumab, durvalumab, and TACE.

Eligibility:

Adults ages 18 and older with intermediate or advanced HCC

Design:

Participants will be screened with a physical exam and medical history. They will have tests to evaluate their hearts as well as blood and urine. A CT and/or MRI scans will be done during the study. If a prior tumor sample is not available; participants may undergo a biopsy. They may undergo an endoscopy of their esophagus and stomach.

Participants will get the study drugs in 21-day cycles:

Two treatment drugs will be injected into a vein every 3 weeks.

Patients will have an interventional treatment procedure done by interventional radiology under sedation; chemotherapy beads will be infused into artery branches in the liver. Participants may have to stay in the hospital for 24 hours for observation, after this procedure. This interventional procedure may be done more than once during the study.

Participants may need to repeat some of the screening tests throughout the study.

Participants may have to stop taking some of their cancer treatment drugs during the study.

Participants will continue on the study until their cancer progresses or until the side effects of the treatment drugs are not tolerable.

DETAILED DESCRIPTION:
Background:

* Worldwide, hepatocellular carcinoma (HCC) is the fourth most common cause of cancer related death with a median survival of 6-9 months.
* Biliary tract carcinoma (BTC) is relatively uncommon and includes cancers of the gallbladder and intra- and extra-hepatic biliary ductal system, although periampullary tumors are often considered part of this group as well.
* A class of agents that in the recent years has been at the epicenter of immunotherapy approaches in gastrointestinal malignancies are the monoclonal antibodies (mAbs) against the immune checkpoint inhibitors CTLA4, PD-1 and PD-L1.
* Durvalumab is a human monoclonal antibody of the immunoglobulin G1 kappa (IgG1 ) subclass. Durvalumab inhibits binding of programmed cell death ligand 1 (PD-L1) to programmed cell death 1 (PD-1) and CD80. Anti-PD-L1 antibodies directly target tumor cells and are expected to have less adverse events in comparison with anti-PD-1 antibodies that target effector T-cells in the tumor microenvironment.
* Tremelimumab is a human IgG2 mAb directed against CTLA-4. Tremelimumab blocks the inhibitory effect of CTLA-4, and therefore enhances T cell activation.
* Angiogenesis is defined as the formation of new blood capillaries, which is a complex process that promotes vascular endothelial growth factor (VEGF) and other proangiogenic factor expression, thus enhancing metastasis. Inhibition of VEGF function by bevacizumab can lead to the inhibition of the new blood vessels formation surrounding a tumor, and consequently arrest the tumor growth by depriving essential nutrients and oxygen.
* TACE has been shown to induce anti-tumor immunity.
* Early phase studies have shown that anti-VEGF treatment with bevacizumab in combination with TACE decreases neovascular formation.
* We have previously shown that locoregional therapies can be safely combined with immune checkpoint blockade. There are also preclinical data suggesting that anti-VEGF therapy may target myeloid cells with suppressor activity.

Objectives:

* To evaluate the 6-month progression free survival (PFS) in participants with advanced HCC BCLC stage B treated with bevacizumab, durvalumab, tremelimumab and TACE.
* To evaluate the 6-month PFS in participants with BTC and HCC BCLC stage C treated with bevacizumab, durvalumab and tremelimumab.
* In participants with BTC enrolled following amendment dated 03/2024, the primary objective will be: To determine if the PFS may be improved upon compared to data from a previous trial in the same participant population.

Eligibility:

* Histopathological confirmation of HCC or BTC or histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of BTC.
* Participants must have evaluable or measurable disease per RECIST 1.1.
* Participants must have disease that is not amenable to potentially curative resection, radiofrequency ablation, or liver transplantation.

Design:

* This is an open label Phase II trial conducted to evaluate efficacy of durvalumab, bevacizumab and tremelimumab combined treatment in participants with advanced HCC BCLC stage C or BTC and efficacy of durvalumab, bevacizumab, tremelimumab and TACE combined treatment in participants with advanced HCC BCLC stage B.
* Initially 3-18 participants with HCC BCLC Stage C or BTC will be enrolled into safety run-in of Arm 1 to determine the safety of combined treatment of durvalumab, bevacizumab and tremelimumab.
* Once safety has been determined, subsequent participants with HCC BCLC Stage C and BTC will be enrolled in Arm 1 and participants with HCC BCLC Stage B will start enrollment into Arm 2, consistent of durvalumab, bevacizumab, tremelimumab and multiple TACE procedures.
* Once Arm 1 has completed accrual in the BTC cohort, Arm 3 will begin accruing participants with advanced unresectable or metastatic BTC, treated with durvalumab, bevacizumab, and tremelimumab using a different treatment schedule.
* Treatment will continue until progression or unbearable toxicity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have

  * histopathological confirmation of HCC (Cohorts 1 and 3)

OR

* histopathological confirmation of BTC or histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of BTC (Cohort 2).

  * Participants should have progressed on standard of care systemic therapy or been intolerant of or have refused standard treatment. Note: For participants enrolled in Cohort 3 (HCC, BCLC stage B), standard of care chemotherapy is not required prior to enrollment.
  * Participants must have disease that is not amenable to potentially curative resection, radiofrequency ablation, or liver transplantation
  * Participants must have evaluable or measurable disease per RECIST 1.1
  * Participants must have at least one lesion accessible for TACE (Cohort 3)
  * Participants must have lesions accessible for biopsy and be willing to undergo pre- and posttreatment biopsies
  * ECOG performance status of 0 to 1
  * If liver cirrhosis is present, patient must have a Child-Pugh score <7
  * Subjects with HCC must have BCLC C (Cohort 1) or BCLC B (Cohort 3)
  * Participants must have normal organ and marrow function as defined below:
* absolute neutrophil count greater than or equal to 1,000/mcL
* platelets greater than or equal to 60,000/mcL
* total bilirubin:if cirrhosis present: Part of Child Pugh requirement-If no cirrhosis: bilirubin should be less than or equal to 2 XULN
* ALT or AST up to 5 x ULN
* Creatinine OR measured or calcutated Creatinine clearance (crCl) (eGFR may Also be used in place of CrCl) A: less than the institutional limit of normal OR greater than or equal to 45/mL/1.73 m^2 for participant with creatinine levels greater than or equal to 1.5 X institutional ULN
* No proteinuria: Urine dipstick <2. Participants discovered to have greater than or equal to 2 + proteinuria on dipstick analysis should undergo a 24-hour urine collection and must demonstrate less than or equal to 1g of protein in 24 hours to be eligible

  * Age greater than or equal to 18 years
  * Participants must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1.
  * The effects of study drugs on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) at the study entry and for the duration of study treatment and up to 90 days after the last dose of the study drug(s). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * HBV infected subjects must be on antivirals and have HBV DNA <100IU/mL. HCV infected subjects can be enrolled with close HCV RNA level monitoring
  * Body weight >30kg
  * Participant must be able to understand and willing to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who have had standard-of-care anti-cancer therapy or therapy with investigational agents (e.g. chemotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies or other investigation agents) or large field radiotherapy within 4 weeks prior to treatment initiation.
* Major surgery within 6 weeks prior to treatment initiation. Minor procedures (e.g. port placement, endoscopy with intervention) within 2 weeks prior to treatment initiation.
* Active central nervous system metastases and/or carcinomatous meningitis. Particpants with known active brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses.
* Medical condition that requires chronic systemic steroid therapy, or any other form of immunosuppressive medication (inhaled and topical steroids are permitted).
* Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID).
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) > 150 mmHg and/or diastolic blood pressure > 100 mmHg), based on an average of 3 BP readings on 2 sessions. Note: anti-hypertensive therapy to achieve these parameters is allowable.
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment
* Evidence of bleeding diathesis or significant coagulopathy (with or without current therapeutic anticoagulation).
* Recent (within 10 days of first dose of study treatment) use of aspirin
* Thromboembolic event within 6 months of initiation of study treatment (including cerebrovascular accident (CVA) and myocardial infarction (MI).
* History of hemoptysis (>2.5 mL of bright red blood per episode) within 1 month prior to treatment initiation.
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* HIV-positive participants are excluded because HIV causes complicated immune deficiency and study treatment can pose more risks for these patients.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Congestive heart failure, transmural myocardial infarction, angina pectoris requiring medication, clinically significant valvular disease, high-risk arrhythmia within 12 months prior to treatment initiation. Prior history of hypertensive crisis or hypertensive encephalopathy.
* Prior invasive malignancies within the past 5 years prior to treatment initiation (with the exception of non-melanoma skin cancers, non-invasive bladder cancer or localized prostate cancer for whom systemic therapy is not required)
* Active or history of inflammatory bowel disease (colitis, Crohn s), irritable bowel disease, celiac disease, or other serious, chronic, gastrointestinal conditions associated with diarrhea.
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to initiation of study treatment.
* History of chronic autoimmune disease (e.g., Addison s disease, multiple sclerosis, Graves disease, Hashimoto s thyroiditis, rheumatoid arthritis, hypophysitis, systemic lupus erythematosus, Wegener s granulomatosis, sarcoidosis syndrome etc.) or other connective tissue diseases with symptomatic disease within the 3 years of initiation of study treatment. Note: Active vitiligo or a history of vitiligo will not be a basis for exclusion.
* Diverticulitis either active or history of within 2 years of initiation of study treatment. Note that diverticulosis is permitted.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that may impair the patient s tolerance of study treatments.
* Received any live vaccine within the last 30 days before treatment initiation.
* Participants who have undergone prior liver transplantation.
* Pregnant women are excluded from this study because durvalumab s and bevacizumab s potential for teratogenic or abortifacient effects is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tremelimumab, durvalumab and bevacizumab, breastfeeding should be discontinued if the mother is treated with study drugs.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the 6-month progression free survival (PFS) in participants with advanced HCC BCLC stage B treated with bevacizumab, durvalumab, tremelimumab and TACE | 6 months
  Proportion of participants with advanced HCC BCLC stage B that have progressive disease after 6 months
To evaluate the 6-month PFS in participants with BTC and HCC BCLC stage C treated with bevacizumab, durvalumab and tremelimumab | 6 months
  Proportion of participants with BTC and HCC BCLC stage C that have progressive disease after 6 months

SECONDARY OUTCOMES:
To determine the best overall response (BOR) rate according to Response Evaluation Criteria (RECIST 1.1) in patients with advanced HCC and BTC | every 9 weeks
  Proportion of patients whose tumors shrunk after therapy
To characterize overall survival (OS) in patients with advanced HCC and BTC treated on this study | death
  Median amount of time subject survives after therapy
To determine the safety and feasibility of bevacizumab, durvalumab, tremelimumab and TACE in patients with advanced HCC | every visit to clinical center
  List of adverse event type, grade and frequency
To determine the safety and feasibility of bevacizumab, durvalumab, tremelimumab in patients with advanced BTC | every visit to clinical center
  List of adverse event type, grade and frequency

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0094.html